CLINICAL TRIAL: NCT02784899
Title: Effect of Iloprost on Pulmonary Oxygenation in Patients With Low Diffusing Capacity During One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2015-0706
Record Dates: First submitted 2016-05-16; First posted 2016-05-27 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Iloprost; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- iloprost group (Experimental): iloprost inhalation group
  Interventions: Drug: iloprost
- control group (Placebo Comparator): normal saline inhalation group
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: iloprost — 20μg(2ml) of inhaled iloprost (Ventavis®)
  When anesthesia induction finishes, change patients' position from supine to lateral position and measure arterial blood gas analysis (ABGA), venous blood gas analysis (VBGA) while two lung is ventilated. After 20 minutes of applying one lung ventilation, measure ABGA. Apply iloprost or normal saline inhalation for each iloprost and control group and measure ABGA at the time of 20 min and 40 min after iloprost (or normal saline) inhalation has finished.
  Arms: iloprost group
Drug: normal saline — 20μg(2ml) of inhaled normal saline
  When anesthesia induction finishes, change patients' position from supine to lateral position and measure ABGA, VBGA while two lung is ventilated. After 20 minutes of applying one lung ventilation, measure ABGA. Apply iloprost or normal saline inhalation for each iloprost and control group and measure ABGA at the time of 20 min and 40 min after iloprost (or normal saline) inhalation has finished.
  Arms: control group

SUMMARY:
One lung ventilation (OLV) is essential during thoracic surgery. During OLV, intrapulmonary shunt can be increased resulting hypoxemia. Although OLV technique had been advanced so far, hypoxemia during OLV reaches about 10% in spite of inspired oxygen fraction 100%. Iloprost is a prostaglandin analogue used for pulmonary hypertension, which can decrease pulmonary artery resistance by selectively dilating pulmonary artery. In this prospective, randomized, double blind study, investigators are planning to investigate the effects of iloprost on respiratory physiology (intrapulmonary shunt, deadspace, oxygenation, etc).

ELIGIBILITY:
Inclusion Criteria:

* scheduled for Video-assisted thoracoscopic surgery (VATS) lobectomy
* 40 < age < 80
* American Society of Anaesthesiologists (ASA) physical status classification I~III
* diffusing capacity (DLCO) <75% at pre op. pulmonary function test

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status classification IV
* New York Heart Association (NYHA) class III~IV
* Severe obstructive lung disease and/or restrictive lung disease patients
* patients with end-organ diseases (i.e. heart failure, respiratory failure, hepatic failure, renal failure)
* arrhythmia
* pregnant women
* disease that can influence the DLCO result (anemia, pulmonary vascular disease)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
PaO2(partial pressure of arterial oxygen) ratio | 40 minutes after iloprost inhalation
incidence of intrapulmonary shunt | 40 minutes after iloprost inhalation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No